CLINICAL TRIAL: NCT01498081
Title: A Randomised, Double-blind, Placebo and Active Controlled, Multi-centre, 6 Way Cross-over, Single-dose Phase IIa Study to Investigate the Local and Systemic Effects of 3 Different Doses of Inhaled AZD2115 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: A Single-dose Study to Investigate the Effects of 3 Different Doses of Inhaled AZD2115 in COPD Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: D3060C00003; EudraCT number: 2011-004641-41
Record Dates: First submitted 2011-12-21; First posted 2011-12-23 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: COPD
Keywords: COPD, pulmonary disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases | interventions — indacaterol; Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (6):
- Single dose of AZD2115 25 µg (Experimental)
  Interventions: Drug: AZD2115
- Single dose of AZD2115 80 µg (Experimental)
  Interventions: Drug: AZD2115
- Single dose of AZD2115 240 µg (Experimental)
  Interventions: Drug: AZD2115
- Single doses of placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Single dose of indacaterol 150 µg (Active Comparator)
  Interventions: Drug: Indacaterol
- Single dose of indacaterol 150 µg + tiotropium 18 µg (Active Comparator)
  Interventions: Drug: Indacaterol + Tiotropium

INTERVENTIONS:
Drug: AZD2115 — AZD2115 administered via inhalation
  Arms: Single dose of AZD2115 240 µg; Single dose of AZD2115 25 µg; Single dose of AZD2115 80 µg
Drug: Placebo — Placebo administered via inhalation
  Arms: Single doses of placebo
Drug: Indacaterol — Indacaterol administered via inhalation
  Arms: Single dose of indacaterol 150 µg
Drug: Indacaterol + Tiotropium — Indacaterol + Tiotropium administered inhalation
  Arms: Single dose of indacaterol 150 µg + tiotropium 18 µg

SUMMARY:
This study in COPD patients will investigate the bronchodilatory effect of AZD2115. AZD2115 will be tested versus placebo and active comparators. The safety and tolerability of AZD2115 including investigations of clinically relevant systemically mediated effects will also be investigated.

DETAILED DESCRIPTION:
A randomised, double-blind, placebo and active controlled, multi-centre, 6 way cross-over, single-dose Phase IIa study to investigate the local and systemic effects of 3 different doses of inhaled AZD2115 in patients with chronic obstructive pulmonary disease (COPD)

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Male or female of non-childbearing potential (post-menopausal or surgically sterilised), age ≥40 years at Visit 1
* Clinical diagnosis of COPD for more than 1 year at Visit 1, according to GOLD guidelines
* Post-bronchodilator FEV1 ≥ 40 to < 80% of the predicted normal value and post-bronchodilator FEV1/FVC < 70%
* Reversible airway obstruction

Exclusion Criteria:

* Significant disease or disorder which, in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the result of the study, or the patient's ability to participate in the study.
* An exacerbation of COPD within 6 weeks prior to Visit 1
* Treatment with systemic glucocorticosteroids with 6 weeks of Visit 2.
* Recent or ongoing respiratory tract infection during enrolment period.
* Need for long-term oxygen therapy and/or saturation O2 < 92%.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-03; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Peak Forced Expiratory Volume in 1 second (FEV1) defined as the maximum FEV1 from the spirometry assessments | During the first 24 hours following administration
Trough FEV1defined as the average FEV1 from the spirometry assessments | During 22 to 26 hours following administration

SECONDARY OUTCOMES:
Average FEV1 | FEV1 0-24h post-dose
Peak, average and trough Forced Vital Capacity (FVC) | FVC peak and average 0-24h post-dose and trough 22-26h post-dose
Systemic effect by assessment of blood pressure (BP) | Peak and average 0-4 h post dose
Systemic effect by assessment of heart rate (HR) and QT interval corrected for heart rate using Fridericia's formula (QTcF) | Peak and average 0-4 h post dose
Systemic effect by assessment of Potassium and Glucose | Peak and average 0-4 h post dose
Safety and tolerability of 3 different single doses of AZD2115 | At screening, during 0-26 h post-dose and at follow-up
Plasma concentrations of AZD2115 after 3 different single doses measured as area under the curve over the time (AUC) and maximum concentration (Cmax), and time to maximum concentration (tmax) | 0-24h post dose

CONTACTS AND LOCATIONS:
Overall Officials: Carin Jorup, MD, Study Director — AstraZeneca R&D Molndal, Sweden
Locations (6):
- Poland (4):
  - Research Site, Bialystok
  - Research Site, Lodz
  - Research Site, Proszowice
  - Research Site, Łęczna
- Sweden (2):
  - Research Site, Gothenburg
  - Research Site, Lund